CLINICAL TRIAL: NCT02164786
Title: Modeling Metabolomic Dynamics Based on Nuclear Magnetic Resonance and High Performance Liquid Chromatography for Severe Patient: a Cohort Study
Brief Title: Metabolomics Dynamics Study for Severe Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: MetaLab_2014_001
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-04

CONDITIONS: Age:18-70 Years; Acute Severe Disease; Acute Physiology And Chronic Health Evaluation(APACHE)II>10
Keywords: Acute severe disease; Intensive care unit; adult; cohort study; metabolomics; NMR; High Performance Liquid Chromatography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma,urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute severe disease

SUMMARY:
Acute severe disease is a major public health challenge that often affects young adults.In past decade, there are lot of new techniques have been developed that aim to improve the outcome of acute severe disease, But few of these works success. According to recently studies, the mortality of the multiple organ dysfunction syndrome（MODS) that is the major cause of death in patients who suffering from acute severe disease, is not improved. On the contrary, if MODS be predicted in early stage of acute severe disease, the death can be prevented. Because acute severe disease poses complex injury that involves multiple pathological processes, understanding the cellular and metabolic network malfunction during acute severe disease is crucial for clinical monitoring and intervention.

Human metabolism is a complex network with hundreds of cross-linked paths. During critical illness, the metabolic network is dynamically disturbed at multiple points. Classical research typically isolates a small part of this network to investigate the impact of pathological physiology molecular mechanisms on clinical outcome. In particular, researchers have examined metabolic disturbances such as cytokine network dysfunction, skeletal muscle breakdown, insulin resistance, dyslipidemia, testosterone and growth hormone/Insulin like growth factor （IGF）dysfunctions, low thyroxine syndrome, and deficiency of vitamin D and calcium with secondary hyperparathyroidism. These complex metabolic disturbances appear and interact at different stages during the pathological process after acute severe illness. Therefore, an integrated approach that combines the biochemical/molecular changes with network disturbances is the key to understanding acute severe illness at the systems biology level and establishing an accurate quantitative model for clinical monitoring.

An interdisciplinary method that includes high-throughput quantitative techniques and effective mathematical and visualization tools is necessary. Furthermore, interdisciplinary methods present the opportunity to develop innovative clinical diagnosis and monitoring methods for severe injuries. The aim of this study is to provide a novel high-throughput method that integrated proton-nuclear magnetic resonance (NMR) metabolomic fingerprinting and High Performance Liquid Chromatography with advance mathematics tools to modeling metabolic dynamics after acute severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-70 years
* Acute Physiology And Chronic Health Evaluation(APACHE)II>10

Exclusion Criteria:

* With comorbidity (Diabetes,Hyperthyroidism or primary organ dysfunction )
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute severe disease
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mortality at hospitalization | Death events from admission to discharge(up to 10 weeks)

SECONDARY OUTCOMES:
Multi Organ Dysfunction Syndrome(MODS) | MODS events occurence from admission to discharge(up to 10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, PhD, MBBS, Study Chair — Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan Academy of Medical Sciences, Chengdu, Sichuan, China